CLINICAL TRIAL: NCT01767571
Title: Open, Two Periods, Two Treatments, Two Sequences, Cross-over, Randomized Study With Single Dosage of Two Oral Preparation of Cephalexin 250 mg/5mL (Ceporex®, GlaxoSmithKline México, S.A. de C.V. vs. Keflex® , Eli Lilly y Compañía de México, S.A. de C.V.) in Fasting Healthy Volunteers
Brief Title: Bioequivalence Study of Cephalexin Suspension 250
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116995
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Infections, Respiratory Tract
Keywords: Mexico; Respiratory infections; Bioequivalence; Cepphalexin
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(reference)/B(test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Cephalexin 125 mg/5ml; Drug: Cephalexin 250mg/5ml
- B(test)/A(reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Cephalexin 125 mg/5ml; Drug: Cephalexin 250mg/5ml

INTERVENTIONS:
Drug: Cephalexin 125 mg/5ml — Reference product 20 ml
  Other Names: Keflex® suspension ELI LILLY Y COMPAÑIA DE MEXICO SA de CV
Drug: Cephalexin 250mg/5ml — Test product 10 ml
  Other Names: Ceporex® suspension GLAXOSMITHKLINE MEXICO SA de CV

SUMMARY:
The objective of this study was to confirm if two formulations of cephalexin suspension are bioequivalent.

Test product was Ceporex® (250 mg Cephalexin / 5 ml; GlaxoSmithKline) and reference product Keflex® (125 mg Cephalexin / 5 ml; Eli Lilly). The single dosage was 10 ml of suspension for Ceporex and 20 ml of suspension for Keflex® .

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fasting conditions.

The population was composed of 28 healthy volunteers, both genders, adults between 18-50 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

Free will participation according to Mexican regulation, Helsinki Declaration, and Good Clinical Practice.

Healthy, between 18 and 50 years. Body Mass Index between 18 and 27.5 In good health by complete medical history and laboratory tests. Blood pressure 130-90/ 90-60 mm Hg; heart rate 55-100 beat per minute, respiratory rate 14-20 movements per minute.

Laboratory tests +/- 10% of normal interval (blood cytology, blood chemistry 27 elements, Hepatitis B and C antigens, HIV, urinalysis, anti-doping, pregnancy, electrocardiogram) -

Exclusion Criteria:

Alteration of vital signs Not complying with inclusion criteria History of cardiovascular, kidney, hepatic, muscular, metabolic, gastrointestinal (including constipation), neurologic, endocrine, hematopoietic (any kind of anemia), asthma, mental or organic disease. Those suffering from muscular trauma 21 days before the beginning of the study.

Requirement of any kind of medication during the course of the study, except study medication.

History of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer. Exposure to medications known as inducers or inhibitors of hepatic enzymes or administration of potentially toxic medication in the 30 days before the study beginning.

Administration of any medication in the 7 half-lives previous to the beginning of the study.

Hospitalization for any cause in the two months before the beginning of the study.

Administration of investigational drugs in the 60 days before the study. Allergy to any medication, food or substance. Alcohol ingestion or intake of beverages containing xanthines (coffee, tea, cocoa, chocolate, mate, cola drinks) or ingestion of charcoal grilled food or grapefruit or orange juice in the 72 hours before the hospitalization or tobacco smoking in the 72 hours before the beginning of the study.

Blood donation or loss => 450 ml in the 60 days before the beginning of the study.

History of drug or alcohol abuse. Special diet requirement, for instance vegetarian diet. Inability to understand nature, aims, and possible consequences of the study. Evidence of non-cooperative attitude during the study. Positive antidoping or pregnancy test Breast-feeding. Females on hormonal treatment.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01-30 (Actual); Primary Completion 2011-02-08 (Actual); Study Completion 2011-02-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of cephalexin | 0.0, 0.083, 0.167, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, and 7.0 postdosage
  Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of cephalexin | 0.0, 0.083, 0.167, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, and 7.0 postdosage
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 116995 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116995?search=study&search_terms=116995#rs